CLINICAL TRIAL: NCT02988011
Title: Influence of Weight Loss by Diet and Surgery on Metabolomic Profile, Body Composition, and Tissue Specific Glucose Uptake: Insights in Type 2 Diabetes Regression (CRUDOS Study)
Brief Title: Improving Glucose and Lipid Metabolism Through Caloric Restriction Using Diet or Surgery (CRUDOS)
Acronym: CRUDOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Ulf Risérus, Associate professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRUDOS AZSciLife
Record Dates: First submitted 2016-12-01; First posted 2016-12-09 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Type2 Diabetes; Weight Loss; Insulin Sensitivity; Metabolism and Nutrition Disorder; Metabolism Disorder, Glucose; Bariatric Surgery Candidate
Keywords: type 2 diabetes; gastric by-pass surgery; low calorie diet; glucose metabolism
MeSH Terms: conditions — Weight Loss; Insulin Resistance; Nutrition Disorders; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2 | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric by-pass surgery (Active Comparator): Gastric by-pass surgery without prior low-caloric diet
  Interventions: Procedure: Gastric by-pass surgery
- Low-caloric diet (Active Comparator): Low-caloric diet followed by gastric by-pass surgery
  Interventions: Procedure: Gastric by-pass surgery; Dietary Supplement: Low-caloric diet

INTERVENTIONS:
Procedure: Gastric by-pass surgery — Gastric by-pass surgery is expected to achieve a mean weight loss of 7-8kg in 4 weeks, which is similar weight-loss achieved in the other arm (low-caloric diet) during this time period.
Dietary Supplement: Low-caloric diet — Energy restricted diet with a total energy intake of 800-1200kcal/day
  Other Names: Energy restricted diet
  Arms: Low-caloric diet

SUMMARY:
In this explorative randomized clinical study, the investigators aim to study metabolic, cellular, and molecular changes that occur during weight loss in obese subjects with and without type 2 diabetes. Using novel "imiomics" (imaging technique using PET/MR bioinformatics) analyses to examine possible metabolic differences between energy restricted diet and gastric by-pass surgery on whole-body and tissue specific insulin sensitivity, glucose tolerance, metabolite and protein profiles, fatty acid metabolism, ectopic fat content, and gene expression in adipose tissue. This study aims to identify novel biomarkers and drug targets for type 2 diabetes as well as validate promising and established biomarkers in an interventional model for improved glucose metabolism.

DETAILED DESCRIPTION:
By using omics platforms such as genomics, proteomics and metabolomics we can have large amount of information about metabolic changes at both tissue and whole body level. In parallel to this, clinical imaging modalities such as Magnetic Resonance Imaging (MRI) and Positron Emission Tomography (PET) have developed rapidly, allowing for whole-body studies of how different tissues are involved in systemic diseases. Furthermore, new hybrid systems such as integrated PET-MRI provide combined information of human morphology and function. The integration of PET with MRI reduces the radiation dose compared with PET-CT to acceptable levels for metabolic studies. To handle the large amounts of data from these examinations we are currently developing an image analysis concept, "Imiomics", that allows holistic analysis of whole-body imaging data with integration of non-imaging data. In the current study, we plan to use PET-MRI as well as imiomics methodology, together with gold standard methodology to assess insulin sensitivity and glucose tolerance in vivo. We aim to conduct a randomized study (CRUDOS study; Caloric Restriction Using Diet Or Surgery) to study glycometabolic effects before and after gastric bypass surgery and low-calorie diet in subjects at different stages of glucose tolerance (i.e. obese subjects with and without T2D).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years
* BMI 35-45
* Sagittal abdominal diameter ≤38.5cm
* For participants with type 2 Diabetes Mellitus, a disease duration of no more than 10 years, treated with 0-3 oral antidiabetic drugs and/or with diet. HbA1C 48-80mmol/mol at baseline visit.

Exclusion Criteria:

* Diabetes complications: proliferative retinopathy, maculopathy, chronic renal failure stadium 3 with an eGFR<60, foot ulcers, symptomatic neuropathy
* Medications within 3 months: Insulin, Thiazolidinediones
* Any other condition with in the opinion of the investigator would render the participant unsuitable for inclusion in the study and /or for the patients safety
* Judgment by the investigator that the subject should not participate in the study if considers subject unlikely to comply with study procedures, restrictions and requirements
* Pregnant or planning to be pregnant during the study.
* Known or suspected history of significant drug abuse.
* History of alcohol abuse or excessive intake of alcohol as judged by investigator.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator
* Sleep apnoea
* Any previous serious cardiovascular event, stroke, acute myocardial infarction.
* Any condition when MRI-PET is contraindicated such as, but not limited to, having a pacemaker or claustrophobia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-02-28 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in tissue specific glucose uptake measured by euglycemic clamp in PET/MR scanner | 4 weeks
  Tissue specific assessment of glucose metabolism (18FDG uptake) using in-scanner (integrated PET-MR) insulin clamps.
Metabolite concentrations in plasma | 4 weeks
  Plasma metabolite concentrations (metabolomics) are assessed by liquid chromatography-mass spectrometry
Gene expression in adipose tissue | 4 weeks
  Change in gene expression is assessed by microarray (untargeted) messenger ribonucleic acid (mRNA) analyses

SECONDARY OUTCOMES:
Lipoprotein changes in plasma assessed by routine clinical chemistry | 4 weeks
Plasma adipokines (e.g. adiponectin) assessed by elisa | 4 weeks
Fatty acid composition in plasma assessed by gas chromatography | 4 weeks
Changes in plasma protein profile (proteomics) assessed by immunohistochemistry | 4 weeks
Epigenetic changes assessed as DNA methylation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Riserus, MMed, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala univeristy hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Most of the data is planned to be shared after the study has ended, the date for when this will occur however needs to be decided.

REFERENCES:
- [Derived] Eriksson JW, Pereira MJ, Kagios C, Kvernby S, Lundstrom E, Fanni G, Lundqvist MH, Carlsson BCL, Sundbom M, Tarai S, Lubberink M, Kullberg J, Riserus U, Ahlstrom H. Short-term effects of obesity surgery versus low-energy diet on body composition and tissue-specific glucose uptake: a randomised clinical study using whole-body integrated 18F-FDG-PET/MRI. Diabetologia. 2024 Jul;67(7):1399-1412. doi: 10.1007/s00125-024-06150-3. Epub 2024 Apr 24. PMID 38656372